CLINICAL TRIAL: NCT03083288
Title: Evaluating in Vivo PARP-1 Expression With 18F-FluorThanatrace Positron Emission Tomography (PET/CT) in Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 26116
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: [18F]FluorThanatrace

INTERVENTIONS:
Drug: [18F]FluorThanatrace — [18F]FluorThanatrace is a radiotracer for PET/CT

SUMMARY:
Up to 30 evaluable participants with known or suspected breast cancer (BIRADS 5 by imaging) will undergo FTT PET/CT imaging before primary surgery or neoadjuvant therapy. Patients undergoing neoadjuvant therapy may choose to have a second FTT PET/CT scan after the start of therapy (1 days to 3 weeks). FTT PET/CT uptake will be correlated with pathology measures and treatment response, in subjects undergoing neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥ 18 years of age
* Known or suspected (BIRADS 5 on imaging) primary breast cancer
* At least one breast lesion one breast lesion that is 1 cm or greater in size by standard imaging (e.g. mammography, ultrasound or breast MRI). Only one type of imaging is required to show a lesion of 1 cm or greater in order for the patient to be eligible to participate in this study. Patients that have a prior diagnosis of primary breast cancer in the opposite breast can be included.
* Willing to allow use orcollection of pathology tissue for the purposes of research from either clinical biopsy or surgical procedure (if adequate tissue is available) or research only biopsy
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McDonald, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald ES, Pantel AR, Shah PD, Farwell MD, Clark AS, Doot RK, Pryma DA, Carlin SD. In vivo visualization of PARP inhibitor pharmacodynamics. JCI Insight. 2021 Apr 22;6(8):e146592. doi: 10.1172/jci.insight.146592. PMID 33884961